CLINICAL TRIAL: NCT02328716
Title: Cytoreduction With or Without Intraoperative Intraperitoneal Hyperthermic Chemotherapy (HIPEC) in Patients With Peritoneal Carcinomatosis From Ovarian Cancer, Fallopian Tube or Primary Peritoneal Carcinoma : Randomized Clinical Trial.
Brief Title: Cytoreduction With or Without Intraoperative Intraperitoneal Hyperthermic Chemotherapy (HIPEC) in Patients With Peritoneal Carcinomatosis From Ovarian Cancer, Fallopian Tube or Primary Peritoneal Carcinoma
Acronym: CARCINOHIPEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EC-GC/AD-01/11; 2011-001715-31 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-31 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Peritoneal Carcinomatosis From Ovarian Cancer; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comparator (Active Comparator): Comparator
  Interventions: Procedure: Cytoreduction
- Experimental (Experimental): Experimental
  Interventions: Procedure: Cytoreduction; Drug: Hipec with Cisplatin

INTERVENTIONS:
Procedure: Cytoreduction — Cytoreduction
Drug: Hipec with Cisplatin — Intraoperative Intraperitoneal Hyperthermic Chemotherapy (Hipec)+Cisplatin
  Arms: Experimental

SUMMARY:
The purpose of this clinical trial is to Investigate whether the administration of HIPEC with Cisplatin (75 milligrams per square meter of body surface) after surgical cytoreduction in women with ovarian, tubal or primary peritoneal carcinoma increased disease-free survival period compared with patients without HIPEC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal carcinomatosis arising from ovarian epithelial carcinoma (stage III or higher), carcinoma of the fallopian tube and primary peritoneal carcinoma.
* Residual tumor < 2.5 mm after completion of cytoreductive surgery.
* Aged < 75 years.
* Baseline ECOG 0-1 (Eastern Cooperative Oncologic Group).
* Adequate bone marrow function with hemoglobin ? 8 g/dl (after correction for iron deficiency anemia), white blood cell count ? 3,000/mm3, platelets ? 100,000/mm3.
* Adequate renal function with creatinine ? 1.5 mg/ dl.
* Adequate liver function with bilirubin levels ? 1.5 mg / dl and AST and ALT ? 80 IU / L.
* Optimal cardiopulmonary function.
* In recurrences, disease-free interval > 6 months.
* Voluntary and signed written informed consent.

Exclusion Criteria:

* Extraperitoneal tumor disease.
* Suboptimal debulking (residual tumor > 2.5 mm).
* Previous history of other malignancies (excluding skin)
* Intestinal obstruction at the time of evaluation.
* Renal failure.
* Heart failure.
* Uncontrolled infection.
* Pregnant or lactating patients.
* In recurrences, disease-free interval < 6 months.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival period | Every 3 months up to 30 months
  Every three months until recurrence of disease.

SECONDARY OUTCOMES:
Evaluation of overall survival. | Every 3 months up to 30 months
  Every three months until recurrence of disease.
Study of morbidity. | Every 3 months up to 30 months
  Every three months until recurrence of disease.
Evaluation of quality of life related to the procedure. | Every 3 months up to 30 months
  Every three months until recurrence of disease.
Study of Ex vivo correlation. | 4 days post surgery
  in vitro cell culture to study the effect of temperature and cisplatin on cell viability

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cascales Campos, M.D Phd, Study Director — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- [Derived] Cascales Campos PA, Gonzalez-Gil A, Gomez-Ruiz AJ, Gil-Gomez E, Alconchel-Gago F, Navarro-Barrios A, Martinez-Garcia J, Alonso-Romero JL, Nieto A, Barcelo-Valcarcel F, Gil-Martinez J. Risk factors and management of incisional hernia after cytoreduction and hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with peritoneal surface malignancies. Hernia. 2020 Apr;24(2):257-263. doi: 10.1007/s10029-019-01962-4. Epub 2019 May 8. PMID 31069579